CLINICAL TRIAL: NCT04541173
Title: A Randomized Phase II Study of Atezolizumab and Bevacizumab With Y-90 TARE in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Brief Title: Study of Atezolizumab and Bevacizumab With Y-90 TARE in Patients With Unresectable Hepatocellular Carcinoma (HCC)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to slow accrual.
Sponsor: Aiwu Ruth He, MD (Other)
Collaborators: Georgetown University (Other); Genentech, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Aiwu Ruth He, MD, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GI19-405
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2024-06-05 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — atezolizumab; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm A (Active Comparator): TARE alone
  Interventions: Other: Y-90 TARE
- Arm B (Experimental): TARE then Bevacizumab and Atezolizumab
  Interventions: Other: Y-90 TARE; Drug: Atezolizumab; Drug: Bevacizumab

INTERVENTIONS:
Other: Y-90 TARE — This plan will involve treating the predominant liver lesions with segment Y-90 TARE using predetermined dosimetry, while keeping FLR equal or greater than 40% (FLR is estimated by excluding the liver volume of Y-90 infused distribution).
  The maximal amount of Y-90 TARE treatment will be limited to only one lobe of the liver if segmental Y-90 TARE is not possible to treat the predominant lesion. Since segmental Y-90 TARE may result in less long term liver damage compared to lobal Y-90 TARE, segmental Y-90 TARE treatment is preferred to lobar Y-90 TARE if segmental Y-90 TARE treatment is able to treat all blood supply to the predominant lesion or lesion with vascular invasion to preserve liver function. For segmental treatment, a minimum tumor dose of 190 Gy should be used for glass microspheres and 120 Gy for resin microspheres. For lobar treatment, a minimum dose of 100 Gy should be used for resin microspheres.
Drug: Atezolizumab — Atezolizumab 1200 mg will be delivered as an IV infusion on Day 1 of each cycle (every 3 weeks). The initial dose will be delivered over 60 (± 15) minutes and if tolerated subsequent infusions may be given over 30 minutes.
  Other Names: Tecentriq
  Arms: Arm B
Drug: Bevacizumab — Bevacizumab 15 mg/kg will be delivered as an IV infusion on Day 1 of each 3 week cycle.The initial dose will be delivered over 90 minutes (±15 minutes) and if tolerated subsequent infusions may be given over 60 minutes
  Other Names: Avastin
  Arms: Arm B

SUMMARY:
This is an open-label, multi-center, randomized phase II study comparing the Y90 TARE followed by bevacizumab and atezolizumab treatment to the Y90 TARE treatment alone in unresectable advanced stage HCC.

DETAILED DESCRIPTION:
Subjects will be randomized to Y-90 TARE alone (Arm A) or Y-90 TARE followed by the combination of atezolizumab and bevacizumab (Arm B). The first 10 subjects randomized to Arm B (Y-90 TARE + bevacizumab + atezolizumab) will be assessed for safety after two cycles. If there are no Grade ≥ 3 unexpected toxicities; possibly, probably or definitely related to TARE in combination with bevacizumab and atezolizumab the combination will be deemed safe and accrual will resume.

Subjects randomized to receive bevacizumab and atezolizumab (Arm B) will start the combination of bevacizumab and atezolizumab 4 weeks (± 1 week) after TARE treatment. Full recovery from the procedure is required prior to systemic treatment:

* AST and ALT ≤ 5 x upper limit of normal (ULN) and total bilirubin ≤ 3 mg/dL
* Manifestations of post-embolization syndrome (e.g., fever, nausea, vomiting, and abdominal pain) have resolved to National Cancer Institute Common Terminology Criteria for Adverse Events, Version 5.0 Grade 1
* No significant medical events (e.g., gastrointestinal [GI] bleeding, cardiac events, hepatorenal syndrome) during or after the TARE procedure.

Arm B subjects will continue the study drugs for a total of 24 months from the TARE treatment, until intolerable toxicity or disease progression occur.

ELIGIBILITY:
Inclusion Criteria:

Subject must meet all of the following applicable inclusion criteria to participate in this study:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately. Patients must be willing and able to provide written informed consent for this trial.
* Age ≥ 18 years at the time of consent.
* ECOG Performance Status of 0-1 at screening
* Histological or cytological evidence/confirmation per AJCC, 8th edition, of hepatocellular carcinoma (HCC).
* Measurable disease by RECIST 1.1.
* Patients must have a Child-Pugh score of A. or selected B7. NOTE: Definition of the selected B7 patients: Child Pugh B7 patients are allowed if they meet the inclusion criteria 11 and they do not have hepatic encephalopathy or more than a moderate amount of ascites.
* Patients must have at least Barcelona Clinic Liver Cancer (BCLC) stage B HCC and must be outside of Milan Criteria; and/or HCC peripheral vascular involvement of any size or number of tumor (segment peripheral, vp1 and vp2 are allowed, but vp3 and vp4 are excluded). NOTE: absence of extrahepatic spread, must be confirmed by computed tomography (CT) or magnetic resonance imaging (MRI) scan of the chest, abdomen, and pelvis.
* Patient must either (1) not be a candidate for liver transplantation as determined by the liver transplant service or (2) refuse evaluation for transplantation.
* Archival tissue obtained within 6 months of registration is required. If archival tissue is not available, subjects are not eligible.
* No prior systemic therapy is permitted. NOTE: Patients who received prior local therapy (e.g., radiofrequency ablation, percutaneous ethanol or acetic acid injection, cryoablation, high-intensity focused ultrasound or TACE) are eligible provided the target lesion(s) have not been previously treated with local therapy or the target lesion(s) within the field of local therapy have subsequently progressed in accordance with RECIST 1.1. Prior TACE is allowed if FLR is ≥ 40%.
* Patient must be a TARE candidate, as defined by a lung dose threshold for Y-90 of 30Gy and an estimated (future liver remnants) FLR of ≥ 40% at the time of forming the comprehensive treatment plan. Both the lung dose threshold and FLR values must be obtained and available in source documentation.
* Patients must demonstrate adequate hepatic, bone marrow, and renal function as defined below. All screening labs should be performed within 14 days of treatment initiation.

  * Hematological

    * Lymphocyte Count: 500/μL
    * Absolute Neutrophil Count (ANC): ≥ 1,500 /μL
    * Hemoglobin (Hgb): ≥ 9 g/dL without transfusion or EPO dependency (within 7 days of assessment)
    * Platelet count (Plt): ≥ 75,000 / μL
  * Renal

    ---Serum creatinine OR Measured or calculated CrCl (GFR can also be used in place of creatinine or CrCl): ≤ 1.5 X upper limit of normal (ULN) OR ≥ 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN
  * Hepatic

    * Bilirubin: ≤ 3.0
    * Aspartate aminotransferase (AST): ≤ 5 X ULN for subjects with cancer in liver
    * Alanine aminotransferase (ALT): ≤ 5 X ULN for subjects with cancer in liver
    * Albumin: > 2.5 mg/dL
    * Urine Protein: Urine dipstick for proteinuria ≤ 2 g (within 14 days prior to initiation of study treatment). Patients discovered to have >2+ proteinuria on dipstick urinalysis at baseline should undergo a 24-hour urine collection and must demonstrate < 1 g of protein in 24 hours.
  * Coagulation

    ---International Normalized Ratio (INR) or Prothrombin Time (PT) Activated Partial Thromboplastin Time (aPTT): ≤ 1.5 X ULN
  * Calcium-Subjects with uncontrolled or symptomatic hypercalcemia are NOT eligible

    * Ionized Calcium: < 1.5 mmol/L
    * Serum Calcium OR Corrected serum calcium: < 12 mg/dL OR < ULN
* Documented virology status of HIV; NOTE: Patients with a positive HIV test at screening are eligible provided they are stable on anti-retroviral therapy, have a CD4 count ≥ 200/µL, and have an undetectable viral load.
* Documented virology status of hepatitis, as confirmed by screening HBV and HCV serology test: For patients with active hepatitis B virus (HBV): HBV DNA <500 IU/mL obtained within 28 days prior to initiation of study treatment, and Anti-HBV treatment (per local standard of care; e.g., entecavir) for a minimum of 14 days prior to study entry and willingness to continue treatment for the length of the study.
* Subjects with chronic infection by HCV who are untreated or who failed previous therapies for HCV are allowed on study. In addition, subjects with successful HCV treatment (defined as sustained virologic response [SVR] 12 or SVR 24) are allowed as long as patients are not actively receiving anti-HCV treatment at the time of study enrollment. Investigators can stop anti-HCV treatment at their discretion prior to enrolling patients on study.
* Females of childbearing potential must have a negative serum pregnancy test within 14 days prior to study treatment. NOTE: Females are considered of child bearing potential unless they are surgically sterile (have undergone a hysterectomy, bilateral tubal ligation, or bilateral oophorectomy) or they are naturally postmenopausal for at least 12 consecutive months.
* Female participants of childbearing potential must be willing to abstain from heterosexual intercourse or to use contraception as outlined in Section 5.6. Male participants capable of fathering children must be willing to abstain from heterosexual intercourse or to use contraception as outlined in Section 5.6.
* As determined by the enrolling physician or protocol designee, ability of the subject to understand and comply with study procedures for the entire length of the study.

Exclusion Criteria

Subjects meeting any of the criteria below may not participate in the study:

* Have signs of liver failure, e.g. clinically significant ascites, encephalopathy, or variceal bleeding within six months from enrollment.
* Uncontrolled pleural effusion, pericardial effusion, or ascites requiring recurrent drainage procedures (once monthly or more frequently). Patients with indwelling catheters (e.g., PleurX® are allowed.
* Untreated or incompletely treated esophageal and/or gastric varices with bleeding or high-risk for bleeding.
* Prior bleeding event due to esophageal and/or gastric varices within 6 months prior to initiation of study treatment. NOTE: Patients must undergo an esophagogastroduodenoscopy (EGD), and all size of varices (small to large) must be assessed and treated per local standard of care prior to enrollment. Patients who have undergone an EGD within 6 months of prior to initiation of study treatment do not need to repeat the procedure.
* Have evidence of excessive hepatopulmonary shunting (> 20% in 99mTc macro-aggregated albumin scan for resin and 30 Gy per treatment for glass) or angiographically demonstrable and non-occludable gastrointestinal shunting, precluding from Y-90 treatment.
* Inadequately controlled arterial hypertension (defined as systolic blood pressure (BP) ≥ 150 mmHg and/or diastolic blood pressure > 100 mmHg), based on an average of ≥ 3 BP readings on ≥ 2 sessions. NOTE: Anti-hypertensive therapy to achieve these parameters is allowable.
* Prior history of hypertensive crisis or hypertensive encephalopathy.
* Significant cardiovascular disease (such as New York Heart Association Class II or greater cardiac disease, myocardial infarction, or cerebrovascular accident) within 3 months prior to initiation of study treatment, unstable arrhythmia, or unstable angina.
* Known fibrolamellar HCC, sarcomatoid HCC, or mixed cholangiocarcinoma and HCC.
* Major surgery within 4 weeks prior to registration or anticipation of a major surgical procedure during study.
* Have had prior transplant of any kind (stem cell or solid organ).
* Have active autoimmune disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids, or immunosuppressive drugs). including, but not limited to, myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis with the following exceptions:

  * Patients with a history of autoimmune-related hypothyroidism who are on thyroid-replacement hormone are eligible for the study.
  * Patients with controlled Type 1 diabetes mellitus who are on an insulin regimen are eligible for the study.
  * Patients with eczema, psoriasis, lichen simplex chronicus, or vitiligo with dermatologic manifestations only (e.g., patients with psoriatic arthritis are excluded) are eligible for the study provided all of following conditions are met:
  * Rash must cover < 10% of body surface area
  * Disease is well controlled at baseline and requires only low-potency topical corticosteroids
  * No occurrence of acute exacerbations of the underlying condition requiring psoralen plus ultraviolet A radiation, methotrexate, retinoids, biologic agents, oral calcineurin inhibitors, or high-potency or oral corticosteroids within the previous 12 months
* Have history of idiopathic pulmonary fibrosis (including bronchiolitis obliterans with organizing pneumonia) drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest CT scan. NOTE: History of radiation pneumonitis in the radiation field (fibrosis) is permitted.
* Treatment with CD137 agonists or immune checkpoint blockade therapies, including anti-CTLA-4, anti-PD-1 and anti-PD-L1 therapeutic antibodies.
* Treatment with systemic immunostimulatory agents (including, but not limited to, interferon and interleukin 2 [IL-2]) within 4 weeks or 5 half-lives of the drug (whichever is longer) prior to initiation of study treatment.
* Treatment with systemic immunosuppressive medication (including, but not limited to, corticosteroids, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-TNF-α agents) within 2 weeks prior to initiation of study treatment, or anticipation of need for systemic immunosuppressive medication during study treatment, with the following exceptions:

  * Patients who received acute, low-dose systemic immunosuppressant medication or a one-time pulse dose of systemic immunosuppressant medication (e.g., 48 hours of corticosteroids for a contrast allergy) are eligible for the study after sponsor-investigator confirmation has been obtained.
  * Patients who received mineralocorticoids (e.g., fludrocortisone), corticosteroids for chronic obstructive pulmonary disease (COPD) or asthma, or low-dose corticosteroids for orthostatic hypotension or adrenal insufficiency are eligible for the study
* Uncontrolled tumor-related pain

  * Patients requiring pain medication must be on a stable regimen at study entry.
  * Symptomatic lesions (e.g., bone metastases or metastases causing nerve impingement) amenable to palliative radiotherapy should be treated prior to enrollment. Patients should be recovered from the effects of radiation. There is no required minimum recovery period.
  * Asymptomatic metastatic lesions that would likely cause functional deficits or intractable pain with further growth (e.g., epidural metastasis that is not currently associated with spinal cord compression) should be considered for loco-regional therapy if appropriate prior to enrollment.
* Patients with brain metastases.
* Have unresolved toxicities from prior anticancer therapy, defined as having not resolved to National Cancer Institute (NCI) CTCAE v5 grade 0 or 1 with the exception of alopecia and laboratory values listed per the inclusion criteria. NOTE: Subjects with irreversible toxicity that is not reasonably expected to be exacerbated by any of the investigational products may be included (e.g., hearing loss) after consultation with the sponsor-investigator.
* Diagnosed or treated for malignancy other than HCC, unless they meet one of the following exceptions:

  * Malignancy treated with curative intent and with no known active disease present for ≥ 2 years before registration and felt to be at low risk for recurrence by the treating physician.
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  * Adequately treated cervical carcinoma in situ without evidence of disease.
* Have a known or suspected allergy to bevacizumab or atezolizumab or known hypersensitivity to Chinese hamster ovary cell products or to any component of the atezolizumab or bevacizumab formulation.
* Significant vascular disease (e.g., aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to initiation of study treatment.
* History of hemoptysis (≥ 2.5 mL of bright red blood per episode) within 1 month prior to initiation of study treatment.
* Evidence of bleeding diathesis or significant coagulopathy (in the absence of therapeutic anticoagulation).
* Current or recent (within 10 days of first dose of study treatment) use of aspirin (≥325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and cilostazol.
* Current or recent (within 10 days prior to study treatment start) use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic (as opposed to prophylactic) purpose. NOTE: Prophylactic anticoagulation for the patency of venous access devices is allowed provided the activity of the agent results in an INR ≤1.5 x ULN and aPTT is within normal limits within 14 days prior to initiation of study treatment.
* Have an uncontrolled intercurrent illness including, but not limited to any of the following:

  * Psychiatric illness/social situations that would limit compliance with study requirements
  * Have any other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that may affect the interpretation of the results or render the patient at high risk from treatment complications.
  * Active alcohol use, drug use, or a psychiatric disease that would, in the opinion of the sponsor-investigator or a sub-investigator (sub-I), prevent the subject from complying with the study protocol and/or endanger the subject during their participation in the study.
* Severe infection within 4 weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia. NOTE: Treatment with therapeutic oral or IV antibiotics within 2 weeks prior to initiation of study treatment Patients receiving prophylactic antibiotics (e.g., to prevent a urinary tract infection or chronic obstructive pulmonary disease exacerbation) are eligible for the study.
* Active tuberculosis.
* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Have received a live attenuated vaccine (e.g., FluMist®) within 30 days of the planned start of study therapy and 180 days after the last dose of the study treatment. NOTE: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however, intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
* Have received or are receiving any investigational therapy within 28 days prior to the first dose of bevacizumab and atezolizumab. NOTE: Subjects may be enrolled in an observational (non-interventional) clinical study or in the follow-up period of an interventional study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2020-11-30 (Actual); Primary Completion 2023-06-18 (Actual); Study Completion 2023-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Aiwu R He, MD, PhD, Principal Investigator — Georgetown University
Locations (6):
- United States (6):
  - Georgetown University, Washington D.C., District of Columbia
  - Moffitt Cancer Center, Tampa, Florida
  - University of Maryland, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Roswell Park Cancer Institute, Buffalo, New York
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: TARE Alone: TARE alone
  Y-90 TARE: This plan will involve treating the predominant liver lesions with segment Y-90 TARE using predetermined dosimetry, while keeping FLR equal or greater than 40% (FLR is estimated by excluding the liver volume of Y-90 infused distribution).
  The maximal amount of Y-90 TARE treatment will be limited to only one lobe of the liver if segmental Y-90 TARE is not possible to treat the predominant lesion. Since segmental Y-90 TARE may result in less long term liver damage compared to lobal Y-90 TARE, segmental Y-90 TARE treatment is preferred to lobar Y-90 TARE if segmental Y-90 TARE treatment is able to treat all blood supply to the predominant lesion or lesion with vascular invasion to preserve liver function. For segmental treatment, a minimum tumor dose of 190 Gy should be used for glass microspheres and 120 Gy for resin microspheres. For lobar treatment, a minimum dose of 100 Gy should be used for resin microspheres.
- Arm B: TARE Then Bevacizumab and Atezolizumab: TARE then Bevacizumab and Atezolizumab
  Y-90 TARE: This plan will involve treating the predominant liver lesions with segment Y-90 TARE using predetermined dosimetry, while keeping FLR equal or greater than 40% (FLR is estimated by excluding the liver volume of Y-90 infused distribution).
  The maximal amount of Y-90 TARE treatment will be limited to only one lobe of the liver if segmental Y-90 TARE is not possible to treat the predominant lesion. Since segmental Y-90 TARE may result in less long term liver damage compared to lobal Y-90 TARE, segmental Y-90 TARE treatment is preferred to lobar Y-90 TARE if segmental Y-90 TARE treatment is able to treat all blood supply to the predominant lesion or lesion with vascular invasion to preserve liver function. For segmental treatment, a minimum tumor dose of 190 Gy should be used for glass microspheres and 120 Gy for resin microspheres. For lobar treatment, a minimum dose of 100 Gy should be used for resin microspheres.
  Atezolizumab: Atezolizumab 1200 mg will be delivered as an IV infusion on Day 1 of each cycle (every 3 weeks). The initial dose will be delivered over 60 (± 15) minutes and if tolerated subsequent infusions may be given over 30 minutes.
  Bevacizumab: Bevacizumab 15 mg/kg will be delivered as an IV infusion on Day 1 of each 3 week cycle.The initial dose will be delivered over 90 minutes (±15 minutes) and if tolerated subsequent infusions may be given over 60 minutes
Period: Overall Study
Arm/Group | Arm A: TARE Alone | Arm B: TARE Then Bevacizumab and Atezolizumab
Started | 3 | 3
Completed | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A: TARE alone
  Y-90 TARE: This plan will involve treating the predominant liver lesions with segment Y-90 TARE using predetermined dosimetry, while keeping FLR equal or greater than 40% (FLR is estimated by excluding the liver volume of Y-90 infused distribution).
  The maximal amount of Y-90 TARE treatment will be limited to only one lobe of the liver if segmental Y-90 TARE is not possible to treat the predominant lesion. Since segmental Y-90 TARE may result in less long term liver damage compared to lobal Y-90 TARE, segmental Y-90 TARE treatment is preferred to lobar Y-90 TARE if segmental Y-90 TARE treatment is able to treat all blood supply to the predominant lesion or lesion with vascular invasion to preserve liver function. For segmental treatment, a minimum tumor dose of 190 Gy should be used for glass microspheres and 120 Gy for resin microspheres. For lobar treatment, a minimum dose of 100 Gy should be used for resin microspheres.
- Arm B: TARE then Bevacizumab and Atezolizumab
  Y-90 TARE: This plan will involve treating the predominant liver lesions with segment Y-90 TARE using predetermined dosimetry, while keeping FLR equal or greater than 40% (FLR is estimated by excluding the liver volume of Y-90 infused distribution).
  The maximal amount of Y-90 TARE treatment will be limited to only one lobe of the liver if segmental Y-90 TARE is not possible to treat the predominant lesion. Since segmental Y-90 TARE may result in less long term liver damage compared to lobal Y-90 TARE, segmental Y-90 TARE treatment is preferred to lobar Y-90 TARE if segmental Y-90 TARE treatment is able to treat all blood supply to the predominant lesion or lesion with vascular invasion to preserve liver function. For segmental treatment, a minimum tumor dose of 190 Gy should be used for glass microspheres and 120 Gy for resin microspheres. For lobar treatment, a minimum dose of 100 Gy should be used for resin microspheres.
  Atezolizumab: Atezolizumab 1200 mg will be delivered as an IV infusion on Day 1 of each cycle (every 3 weeks). The initial dose will be delivered over 60 (± 15) minutes and if tolerated subsequent infusions may be given over 30 minutes.
  Bevacizumab: Bevacizumab 15 mg/kg will be delivered as an IV infusion on Day 1 of each 3 week cycle.The initial dose will be delivered over 90 minutes (±15 minutes) and if tolerated subsequent infusions may be given over 60 minutes
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Continuous [Median (Full Range); unit: years] | 72 [59 to 82] | 72 [67 to 75] | 72 [59 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 3
  Male | 1 | 2 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 1 | 2
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
ECOG Performance Status [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) from 0-5 that describes a patient's level of functioning where 0=Fully active, able to carry on all pre-disease performance without restriction, 1 = Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature, e.g., light house work, office work and 5=Dead.
  Participants
    ECOG = 0 | 1 | 1 | 2
    ECOG = 1 | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS) by RECIST 1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  PFS is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Up to a maximum of 16 months.
Population: Due to the early termination of the study by the funder and sponsor-investigator, pre-planned analyses were not conducted. In lieu of this analysis, the raw response data per RECIST 1.1 is presented per-arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 3 | 3
Participants
  Stable Disease per RECIST 1.1 (SD) | 2 | 0
  Partial Response per RECIST 1.1 (PR) | 0 | 1
  Progressive Disease per RECIST 1.1 (PD) | 1 | 2

2. Secondary Outcome: Adverse Events
Description: Number of subjects experienced toxicity per Common Terminology Criteria for Adverse Events (CTCAE) v5.
Time Frame: 14 months
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 3 | 3
Participants | 2 | 3

3. Secondary Outcome: Progression Free Survival by mRECIST
Description: Per modified RECIST (mRECIST), Complete Response (CR), the disappearance of any intratumoral arterial enhancement in all target lesions; Partial response(PR), >= 30% decrease in the sum of diameters of viable (contrast enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions; Progressive disease(PD), >= 20% increase in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since the treatment started; Stable disease(SD), any cases that do not qualify for either partial response or progressive disease.
  PFS is defined as the time from randomization to the first occurrence of disease progression or death from any cause (whichever occurs first) according to mRECIST
Time Frame: Up to a maximum of 16 months.
Population: Due to the early termination of the study by the funder and sponsor-investigator, pre-planned analyses were not conducted. In lieu of this analysis, the raw response data per mRECIST is presented per-arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 3 | 3
Participants
  Partial Response per mRECIST (PR) | 0 | 1
  Stable Disease per mRECIST (SD) | 2 | 0
  Progressive Disease per mRECIST (PD) | 1 | 2

4. Secondary Outcome: Time to Progression (TTP) by mRECIST
Description: Per modified RECIST (mRECIST), Complete Response (CR), the disappearance of any intratumoral arterial enhancement in all target lesions; Partial response(PR), >= 30% decrease in the sum of diameters of viable (contrast enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions; Progressive disease(PD), >= 20% increase in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since the treatment started; Stable disease(SD), any cases that do not qualify for either partial response or progressive disease.
  TTP is defined as the time from randomization to the first occurrence of disease progression according to mRECIST
Time Frame: Up to a maximum of 16 months.
Population: Due to the early termination of the study by the funder and sponsor-investigator, pre-planned analyses were not conducted. In lieu of this analysis, numerical median of TTP is presented per-arm.
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 3 | 3
Months | 12.71 [8.67 to 12.71] | 11.96 [5.78 to 15.18]

5. Secondary Outcome: Overall Response Rate (ORR) by mRECIST
Description: Per modified RECIST (mRECIST), Complete Response (CR), the disappearance of any intratumoral arterial enhancement in all target lesions; Partial response(PR), >= 30% decrease in the sum of diameters of viable (contrast enhancement in the arterial phase) target lesions, taking as reference the baseline sum of the diameters of target lesions; Progressive disease(PD), >= 20% increase in the sum of the diameters of viable (enhancing) target lesions, taking as reference the smallest sum of the diameters of viable (enhancing) target lesions recorded since the treatment started; Stable disease(SD), any cases that do not qualify for either partial response or progressive disease.
  ORR is defined as a complete or partial response according to mRECIST
Time Frame: Up to a maximum of 16 months
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 3 | 3
Participants
  Complete Response per mRECIST (CR) | 0 | 2
  Partial Response per mRECIST (PR) | 2 | 0
  Stable Disease per mRECIST(SD) | 1 | 1

6. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to death from any cause.
Time Frame: Upto a maximum of 18 months
Population: Due to the early termination of the study by the funder and sponsor-investigator, pre-planned analyses were not conducted. In lieu of this analysis, the survival status is presented per-arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 3 | 3
Participants
  Alive | 3 | 3
  Expired | 0 | 0

7. Secondary Outcome: Subject Function
Description: Patient-reported outcomes (PRO) instrument is a reduced version of the European Organisation for Research and Treatment of Cancer (EORTC QLQ-C30) which includes only questions related to the physical, role, emotional, and social function domains, as well as overall health-related quality of life. All of the scales measures range in score from 0 to 100. A high score for a functional scale represents a high / healthy level of functioning (a score of 100 indicates a good health status and a score of 0 indicates severe impairments). A high score for the global health status / QoL represents a high QoL. If items I1, I2, ... In are included in a scale, the procedure is as follows: RawScore = RS = (I1 + I2+…. + In)/n; Apply the linear transformation to 0-100 to obtain the score S, Functional scales: S = {1 - ((RS-1)/range)}*100; QoL: S = {(RS-1)/range}*100; Range is the difference between maximum and minimum possible value of RS. Subject function will be assessed via PRO instrument.
Time Frame: 16 months
Population: Due to the early termination of the study by the funder and sponsor-investigator, pre-planned analyses were not conducted. In lieu of this analysis, the mean scores at baseline for each function are presented per-arm. Scores were not available for 1 subject in Arm A and 1 subject in ARM B.
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 2 | 2
score on a scale
  Physical functioning | 70 [60 to 80] | 93.33 [86.67 to 100]
  Role functioning | 91.67 [83.33 to 100] | 50 [0 to 100]
  Emotional functioning | 75 [66.67 to 83.33] | 70.83 [66.67 to 75]
  Social functioning | 91.67 [83.33 to 100] | 91.67 [83.33 to 100]
  QoL | 70.83 [50 to 91.67] | 79.17 [75 to 83.33]

8. Secondary Outcome: Overall Response Rate (ORR) by RECIST1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR is defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1.
Time Frame: Up to a maximum of 16 months
Population: Due to the early termination of the study by the funder and sponsor-investigator, pre-planned analyses were not conducted. In lieu of this analysis, the raw response data per RECIST1.1 is presented per-arm.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 3 | 3
Participants
  Complete Response per RECIST1.1 (CR) | 0 | 1
  Partial Response per RECIST1.1 (PR) | 1 | 0
  Stable Disease per RECIST1.1 (SD) | 2 | 2

9. Secondary Outcome: Time to Progression (TTP) by RECIST1.1
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  TTP is defined as the time from randomization to the first occurrence of disease progression according to RECIST v1.1
Time Frame: Up to a maximum of 16 months.
Population: as for outcome 4
Measure: Median (Full Range); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 3 | 3
Months | 12.71 [8.67 to 12.71] | 11.96 [5.78 to 15.18]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 18 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 14 months.
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 1/3 | 0/3
Other Adverse Events (participants affected / at risk) | 2/3 | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=3) | Arm B (N=3)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=3) | Arm B (N=3)
FATIGUE (General disorders) | 2 (3) | 3 (9)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 1 (1) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
CHILLS (General disorders) | 0 (0) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 0 (0) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 2 (8)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 1 (5)
POSTNASAL DRIP (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
VOMITING (Gastrointestinal disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-12-02): https://cdn.clinicaltrials.gov/large-docs/73/NCT04541173/Prot_SAP_000.pdf